CLINICAL TRIAL: NCT01568242
Title: Changes in Vitreous Temperature During Phacoemulsification
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APEC-VitTemp
Record Dates: First submitted 2012-02-23; First posted 2012-04-02 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Cataract; Phacoemulsification; Temperature; Vitreous
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thermoprobe (Experimental): Determination of vitreous temperature with a thermoprobe
  Interventions: Device: Phacoemlsification

INTERVENTIONS:
Device: Phacoemlsification — Transurgical measurement of temperature
  Other Names: Thermoprobe

SUMMARY:
Temperature in the vitreous cavity decreases during vitrectomy, and the same effect is seen during an uneventful phaco surgery. Significant changes occur between the baseline temperature and after every step of the surgery.

DETAILED DESCRIPTION:
A 23-gauge thermometer probe inserted prior to the beginning of the cataract surgery to measure the vitreous temperature at different stages of the procedure (capsulorrhexis, hydrodissection, phacomulsification, irrigation/aspiration and intraocular lens (IOL) implantation). Room temperature also registered during every step. At the end of the surgery, oral temperature will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the Retina department that underwent phacoemulsification and vitrectomy

Exclusion Criteria:

* Posterior capsule rupture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Vitreous temperature | Every five minutes during a phacoemulsification procedure, and at every step of the surgery
  Temperature of the vitreous is taken every five minutes from the start of a phacoemulsification. Also Temperature is take after every step of the surgery (capsulorhexis, hydrodissection, phacoemulsification, irrigation/aspiration, IOL implantation).

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz-Mercado, MD, Study Chair — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación Para Evitar la Ceguera en México, Mexico City, Mexico City, Mexico